CLINICAL TRIAL: NCT04624672
Title: GLP-1 Agonists as Neoadjuvant Therapy for Surgical Treatment of Type 2 Diabetes: A Randomized Controlled Trial
Brief Title: Treatment of GLP-1 for Diabetic Bariatric Patients
Acronym: NOVO-GLP1
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Geisinger Clinic (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Christopher Still, Director of Obesity Institute, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-0937; U1111-1242-4068 (Other: NOVO Nordisk)
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Bariatric Surgery; Semaglutide
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Arm (Placebo Comparator): Once weekly injection of placebo 4-6 months at prescribed dose
  Interventions: Drug: Placebo
- Test Arm (Active Comparator): Once weekly injection of 1.0mg Semaglutide 4-6 months at prescribed dose
  Interventions: Drug: Semaglutide (1 Mg Dose)

INTERVENTIONS:
Drug: Semaglutide (1 Mg Dose) — Weekly injection of study drug for 4-6 months prior to Roux-en-Y gastric bypass surgery
  Other Names: semaglutide
  Arms: Test Arm
Drug: Placebo — Weekly injection of placebo for 4-6 months prior to Roux-en-Y gastric bypass surgery
  Arms: Control Arm

SUMMARY:
This study is for patients that are diabetic, and require insulin for glycemic control, and going through the bariatric surgery process. This is a prospective study that is trying to determine if the introduction of a semaglutide increases the remission rates of diabetes post-operatively.

DETAILED DESCRIPTION:
The evidence to date supporting the association between treatment with GLP-1 agonists and diabetes remission after metabolic surgery is based on retrospective studies. This study is a 2:1 randomized, blinded, parallel, prospective placebo-controlled trial with a standardized treatment approach in order to establish the role of GLP-1 in remission of diabetes after metabolic surgery. This study will enroll 126 patients, with the goal of 100 patients completing the clinical trial (33 in the Placebo/Control Group and 67 in the Test Group).

The preoperative program for Metabolic Surgery involves multidisciplinary health evaluation and care, as well as patient education lasting approximately 6 months. Patients that consent to the clinical trial, will receive study drug on top of the standard care that is provided for 4 months prior to bariatric surgery. During this time, glycemic control will be monitored carefully through points of contact with the study team and additional lab assessments for the clinical trial. After bariatric surgery, patients will continue in the study for 2 years and glycemic control will be managed according to the current standard of care for perioperative glucose control. During this time, patients will continue to meet with the study team and collect lab assessments

All study patients will be followed for two years after metabolic surgery. Efficacy and outcomes will be evaluated by comparative analysis of laboratory results (Labs 1-6) which monitor longitudinal glycemic control. Outcomes will then be compared between Test and Control groups. The major study outcomes will be diabetes remission as defined by the American Diabetes Association. Secondary outcomes will include measures of improvement in glycemic control and beta cell function (change in fasting glucose levels, HbA1C, and C- peptide). All study labs and chemistry analysis will be performed at the Geisinger Medical Laboratory which is accredited by the College of American Pathologists and the Centers for Medicare and Medicaid - Clinical Laboratory Improvement Amendments (CLIA) and licensed by the Pennsylvania Department of Health Division of Laboratories. Evaluation of the continued need for medications for diabetes treatment will be the responsibility of the study team. Longitudinal information relating to medication use will be derived from direct patient contact at study visits, and review of standard of care medicine reconciliations from the Electronic Health Record.

ELIGIBILITY:
Inclusion Criteria:

1. Candidates for Roux-en-Y Gastric Bypass Surgery with an established diagnosis of Type 2 diabetes requiring insulin treatment for glycemic control
2. Ability to provide informed consent before any trial-related activities

Exclusion Criteria:

1. Prior metabolic surgery procedure
2. Use of GLP-1 analogues for diabetes treatment at the time of recruitment
3. Known or suspected allergy to semaglutide or the excipients in semaglutide, or related products.
4. Contraindications to semaglutide which include a personal or family history of medullary carcinoma of the thyroid or multiple endocrine neoplasia syndrome-2 (MEN-2)
5. Previously randomized for participation in this trial.
6. Pregnant, breast-feeding or the intention of becoming pregnant or not using adequate contraceptive measures.
7. Type 1 diabetes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Still, DO, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Medical Center, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Arm | Test Arm
Started | 2 | 1
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — Early Study Closure | 2 | 1

BASELINE CHARACTERISTICS:
Population: Due to low recruitment numbers (>5), no data analysis was completed because total number of patients recruited is too low to ensure patient confidentiality.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Test Arm | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment

OUTCOME MEASURES:

1. Primary Outcome: RATE OF PARTIAL REMISSION OF DIABETES
Description: HbA1C < 6.5%, fasting glucose <125 mg/dl, or no medications or active treatment for one year
Time Frame: 11 months
Population: as for baseline characteristics
Arm/Group | Control Arm | Test Arm
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: RATE OF COMPLETE REMISSION OF DIABETES
Description: HbA1C < 6.0%, fasting glucose <100 mg/dl, or no medications or active treatment for o
Time Frame: 11 months
Population: as for baseline characteristics
Arm/Group | Control Arm | Test Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Control Arm | Test Arm
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/72/NCT04624672/Prot_SAP_000.pdf